CLINICAL TRIAL: NCT05994183
Title: The Bronchiolitis in Hospitalized Infants (BroncHI) Study: A Feasibility Trial Aimed to Identify and Treat Hospitalized Infants With Bronchiolitis Most at Risk for Recurrent Wheezing and Asthma
Brief Title: The Bronchiolitis in Hospitalized Infants Study
Acronym: BroncHI
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was withdrawn with no participants enrolled due to the need for an IND from the FDA, which significantly expanded the scope of the study beyond what was originally anticipated for a pilot project within this network.
Sponsor: IDeA States Pediatric Clinical Trials Network (Network)
Collaborators: National Institutes of Health (NIH) (NIH); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 275605
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Bronchiolitis
Keywords: Infants <24 months of age hospitalized with bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: An open-label single-arm pilot study to assess feasibility of study procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexamethasone Administration (Experimental): Dexamethasone will be given orally to all consented participants. Two doses will be administered within 12-48 hours, with at least the 1st dose administered during the bronchiolitis hospitalization. If the participant is discharged before the 2nd dose, it will be administered at home.
  Interventions: Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Dexamethasone Oral — Dexamethasone 0.6 mg/kg/dose orally (max 16 mg/dose)

SUMMARY:
The goal of this clinical trial is to determine whether it is possible to identify, enroll, and deliver the study intervention (the corticosteroid dexamethasone) in hospitalized infants with bronchiolitis.

Participants in this study will be given two doses of dexamethasone within 72 hours of enrollment, followed by 30 days of safety monitoring.

Results of this feasibility pilot study may be used to inform the design of a future randomized controlled trial, whose results in turn could induce a paradigm shift in acute management of bronchiolitis.

DETAILED DESCRIPTION:
This is a open-label single-arm pilot study to assess feasibility of study procedures. The study population is infants <24 months of age, admitted with a physician diagnosis of non-RSV bronchiolitis that meet at least one of the following criteria: 1) history of breathing problems, 2) history of eczema, and/or 3) family history of asthma.

The primary objective is to assess the ability to administer 2 doses of dexamethasone to infants hospitalized with bronchiolitis meeting the inclusion criteria. The literature suggests that prompt intervention in the course of bronchiolitis disease is important for possibly altering the immune response and sequelae. Therefore, it is important that we are able to demonstrate the ability to initiate the intervention while the child is still hospitalized and complete the number of doses with the desired anti-inflammatory effect. We aim to successfully administer both doses of the study medication in 87% of infants enrolled.

Enrolling sites will recruit participants in collaboration with outpatient practices within Environmental influences on Child Health Outcomes (ECHO) Institutional Development Award (IDeA) States Pediatric Clinical Trials Network (ISPCTN) states that provide primary care services to children (<24 months old). Sites will serve a population base of at least 40% Medicaid/uninsured children, <60% non-Hispanic White children, or >40% of families residing in rural communities.

Participants will be enrolled on the study for approximately 30 days. While in the study they will receive dexamethasone at a dose of 0.6 mg/kg/dose orally (max 16 mg/dose) per day for 2 days. The 1st dose will be given while the infant is inpatient (within 24 hours following enrollment). The 2nd dose will be given on Day 2, either inpatient or at home. The time interval between doses will be between 12 and 48 hours. Participants will be followed for safety information 30 days (±4 days) after the 2nd dose.

The study duration is 24 months (2 months start-up, 17 months enrollment, 1 month follow-up, and 3 months close-out and data analysis).

ELIGIBILITY:
Inclusion Criteria:

* Infants <24 months of age at time of enrollment
* Admitted to the hospitalist service with a diagnosis of bronchiolitis
* RSV and COVID-19 Negative
* At least one of the following clinical criteria:

  * personal history of breathing problems
  * personal history of eczema
  * parental history of asthma
* Parental ability to speak and read English or Spanish

Exclusion Criteria:

* Preterm Infant (born at < 34 weeks' gestation)
* Diagnosis of asthma
* Known underlying heart failure, hypertension, gastrointestinal bleeding, liver disease, thyroid disease (per parental report and chart review)
* Currently taking corticosteroids (inhaled or oral) or have taken corticosteroids within 7 days prior to hospitalization (per parental report and chart review)
* Admission to the intensive care unit (ICU) at time of enrollment
* Participants (caregivers) who, in the view of the investigator, whom are unlikely able to comply with the protocol requirements

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2025-03-09 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants that receive 2 doses of dexamethasone per protocol. | Intervention: 72 hours; Follow-up: 30 days
  A total of N=30 recruited participants will be enrolled into the study. In the primary objective, we expect 26 out of 30 (87%) participating infants will successfully receive 2 doses of dexamethasone per protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Neemann, MD, Study Chair — University of Nebraska; Ashley Deschamp, MD,MS, Study Chair — University of Nebraska
Locations (2):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
The study team will place participant's de-identified data and other limited information, such as race and ethnic group, into one or more centralized database(s). The study team will share this data in compliance with the ISPCTN and NIH data sharing policies.
Supporting Information: SAP
Time Frame: NIH Public Access Policy ensures public access to the published results of NIH-funded research. Scientists are required to submit final peer-reviewed journal manuscripts from NIH funds to the digital archive PubMed Central upon publication acceptance.
  ECHO ISPCTN Publications and Presentations Policy, ensures accurate, responsible, and efficient communication of findings from ECHO ISPCTN clinical trials. The ECHO ISPCTN Steering Committee has approved and ratified the Publications and Presentations Policy, which includes representatives from all site awardees, as well as representatives from NIH and the DCOC NIH Data Sharing Policy, the policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission Rule. Trial results will be submitted to ClinicalTrials.gov. Additional plans are to publish results in peer reviewed journals. Researchers may request trial data by contacting Jeannette Lee, PhD, at the DCOC.
Access Criteria: TBA